CLINICAL TRIAL: NCT06592495
Title: Bioepuivalence Study for the Safety and the Pharmacokinetics of DWJ1589 and DWC202315 in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Bioepuivalence Study for the Safety and the Pharmacokinetics of DWJ1589 and DWC202315
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1589101
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: RTRT (Experimental): T: DWJ1589 R: DWC202315
  Interventions: Drug: Period 1; Drug: Period 2; Drug: Period 3; Drug: Period 4
- Sequence B: TRTR (Experimental): T: DWJ1589 R: DWC202315
  Interventions: Drug: Period 1; Drug: Period 2; Drug: Period 3; Drug: Period 4

INTERVENTIONS:
Drug: Period 1 — DWJ1589 or DWC202315
Drug: Period 2 — DWJ1589 or DWC202315
Drug: Period 3 — DWJ1589 or DWC202315
Drug: Period 4 — DWJ1589 or DWC202315

SUMMARY:
This study aims to evaluate the safety and pharmacokinetic characteristics after administration of DWJ1589 and DWC202315 in healty adult volunteers.

DETAILED DESCRIPTION:
The study design is a Randomized, Open-label, Oral, Single-dose, 2 × 4 crossover study. The patients were randomly assigned to each group. Primary endpoint was Cmax and AUClast of DWJ1589 and DWC202315. Secondary endpoints were AUCinf, AUClast/AUCinf, Tmax and t1/2 of DWJ1589 and DWC202315.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 year old
* Healthy adult volunteers

Exclusion Criteria:

* with a history of mental disorder
* For female volunteers, those who are suspected of being pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The maximum serum concentration(Cmax) of DWJ1589 and DWC202315 | At pre-dose (0 hour), and post-dose 0.83 to 72 hour.
  Cmax of DWJ1589 and DWC202315
The Area under the curve(AUC)last of DWJ1589 and DWC202315 | At pre-dose (0 hour), and post-dose 0.83 to 72 hour.
  AUClast of DWJ1589 and DWC202315

CONTACTS AND LOCATIONS:
Overall Officials: KANG, MD, PhD, Principal Investigator — H Plus Yangji Hospital

IPD SHARING:
Plan to Share IPD: No